CLINICAL TRIAL: NCT04392505
Title: Durvalumab (MEDI4736) After chemoRadioTherapy (DART) for NSCLC Patients - a Phase II Translational and Biomarker Study Investigating PDL1 Positive and Negative Patients
Brief Title: Durvalumab(MEDI4736) After chemoRadioTherapy(DART) for NSCLC-a Translational and Biomarker Study
Acronym: DART
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Åslaug Helland, Prof, MD, Head of Research, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DART
Record Dates: First submitted 2020-05-08; First posted 2020-05-19 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cancer; Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Stage III; NSCLC; NSCLC, Stage III
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: open, exploratory, multinational, phase 2 trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The whole study population (Experimental): All patients will receive durvalumab for up to 1 months after standard treatment With chemoradiotherapy.
  Interventions: Drug: Durvalumab Injection

INTERVENTIONS:
Drug: Durvalumab Injection — Included patients will receive durvalumab (fixed dose, 1500mg Q4W) until progressive disease and no clinical benefit, intolerable toxicity or patient's wish, for a maximum duration of 12 months. Treatment with durvalumab should start <5 weeks after last radiotherapy dosing.
  Other Names: Imfinzi

SUMMARY:
The main aim is to identify and describe biomarkers in different sample types related to chemoradiation followed by durvalumab treatment for stage III PD-L1 negative and positive non-small cell lung cancer (NSCLC) patients' eligible for curatively intended chemoradiation.

The hypothesis is that clinical differences in course of disease reflect underlying biological characteristics.

DETAILED DESCRIPTION:
This is an open, multinational, phase 2 trial to investigate the Properties of cancer cells before, during and after treatment with the investigational study drug durvalumab in patients with locally advanced non-small celled lung cancer (NSCLC). Both patients with high and low PD-L1 expression are allowed to participate. Durvalumab (PD-L1 inhibitor) will be administered after a period with standardtreatment with chemotherapy and radiationtherapy (chemoradiotherapy) for around 7 weeks. After maximum 5 weeks break after chemoradiotherapy, durvalumab will be given in the same dose to all patients for up to 12 months. The follow-up include a safety follow-up for up to five years, followed by a survival follow-up for up to a total of ten years.

The main aim is to identify and describe biomarkers in different sample types related to chemoradiation followed by durvalumab treatment for stage III PD-L1 negative and positive non-small cell lung cancer (NSCLC) patients' eligible for curatively intended chemoradiation.

The hypothesis is that clinical differences in course of disease reflect underlying biological characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Locally-advanced, unresectable, stage III NSCLC (including PET-CT and MRI-brain in the diagnostic work-up).
2. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
3. Diagnostic biopsy with PD-L1 <1% in 50 patients PD-L1 ≥1% in 50 patients
4. Adequate core or excisional biopsy for tumor assessment
5. Age > 18 years at time of study entry
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Life expectancy of at least 12 weeks
8. Body weight >30 kg
9. Adequate normal organ and marrow function as defined below:

   - Haemoglobin ≥9.0 g/dL
   * Absolute neutrophil count (ANC) 1.5 x (> 1500 per mm3)
   * Platelet count ≥100 x 109/L (>75,000 per mm3)
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN).
   * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
   * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   - Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

   Females:

   - Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
10. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
11. Women of childbearing potential (WOCBP) should have a negative urine or serum pregnancy within 7 days prior to receiving the firs dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. A woman is considered as WOCBP, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
12. WOCBP should use an adequate method to avoid pregnancy
13. males who are sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for a period of 90 days (duration of sperm turnover) / the time required for the investigational drug to undergo five half-lives
14. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Non-small cell lung cancer disease suitable for curative surgery
2. Significant cardiac, pulmonary or other medical illness that would limit activity or survival
3. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study during the last 2 weeks.
4. Any concurrent chemotherapy, Investigational Product (IP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
5. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
6. History of allogenic organ transplantation.
7. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stableon hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone

i. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent j. History of another primary malignancy except for

* Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ without evidence of disease k. History of active primary immunodeficiency or medical condition requiring high doses (>30 mg prednisolone daily) of systemic steroids or other forms of immunosuppressive therapy l. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), and hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

  m. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:
* Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
* Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.

  n. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.

  o. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

  p. Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.

  q. Judgement by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

  r. Patients with grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study physician.

  s. Patients with irreverible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consulation with the Study Physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2033-05-01 (Estimated)

PRIMARY OUTCOMES:
Impact of tumour mutational burden (TMB) measured in the tumour tissue and blood samples, on the hazard. | Throughout study, up to 5 years
  Analyses of TMB in tumour tissue. Patients with high Tumour Mutational Burden, TMB (> 8.5 mutations per megabase) have a hazard ratio equal to or less than 0.55 as compared to patients with low TMB. Tumor tissue will be analysed in regard to TMB, and several different cut-offs will be evaluated.

SECONDARY OUTCOMES:
Predict assosiation between Tumour Mutational Burden, TMB, measured in tumour tissue and blood samples and clinical response | Through study, up to 5 years
  To investigate different levels of TMB in tumor tissue compared to blood samples, as predictors for development of clinical response
Specific RNA profiles predict response to treatment | Through study, up to 5 years
  Transcriptome characterization (RNA-sequencing) on tumour material to investigate this
Impact of Molecular profiles in urine on response to treatment | Through study, up to 5 years
  To investigate urine for predictive biomarkers (ctDNA, miRNA)
Analysis of pre-treatment and under-treatment samples may identify biomarkers for predicting which patients will benefit from treatment with durvalumab after chemoradiation | Through study, up to 5 years
  Analyses of biomarkers in tumour tissue.
The durvalumab treatment following chemoradiation will induce T cell responses against antigens expressed in each patient´s tumor. | Through study, up to 5 years
  Immunological response assessment performed on tumour material from participants.
A possible change in PD-L1 status will be explored | Through study, up to 5 years
  Immunohistochemistry of PD-L1 assessed on tumour tissue.
The durvalumab treatment following chemoradiation has acceptable safety and tolerability in NSCLC patients, as assessed by Patient Reported Outcome measurements. | Through study, up to 5 years
  Patient reported outcome measurements by standardized Tools; EORTC-QLQ-C30 and LC13.

OTHER OUTCOMES:
The gut microbiome influence the responses to chemoradiation followed by durvalumab | Through study, up to 5 years
  Genetic analyses on feces samples, by use of feces "Cards".

CONTACTS AND LOCATIONS:
Overall Officials: Åslaug Helland, Prof, MD, Principal Investigator — Oslo University Hospital
Locations (10):
- North Estonia Medical Centre, Tallinn, Estonia
- Finland (3):
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- National Cancer Institute, Vilnius, Lithuania
- Norway (5):
  - Haukeland universitetssykehus, Bergen
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - Universitetssykehuset i Nord-Norge, Tromsø
  - St. Olavs Hospital, Trondheim

REFERENCES:
- [Derived] Horndalsveen H, Haakensen VD, Madebo T, Gronberg BH, Halvorsen TO, Koivunen J, Oselin K, Cicenas S, Helbekkmo N, Aanerud M, Ahvonen J, Silvoniemi M, Bjaanaes MM, Farooqi S, Nebdal D, Dalsgaard AM, Danielsen BK, Borve M, Dalen TS, Ojlert AK, Helland A. Blood-based tumor mutational burden as a biomarker in unresectable non-small cell lung cancer treated with chemoradiotherapy and durvalumab. Front Oncol. 2025 Oct 22;15:1681420. doi: 10.3389/fonc.2025.1681420. eCollection 2025. PMID 41199847
- [Derived] Langberg CW, Horndalsveen H, Helland A, Haakensen VD. Factors associated with failure to start consolidation durvalumab after definitive chemoradiation for locally advanced NSCLC. Front Oncol. 2023 Jul 5;13:1217424. doi: 10.3389/fonc.2023.1217424. eCollection 2023. PMID 37476372